CLINICAL TRIAL: NCT07247409
Title: Establishment of Hong Kong Diabesity Register
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Alice Pik Shan KONG, Professor, Chinese University of Hong Kong
Other Study IDs: CRE 2025.324 register
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Diabesity
MeSH Terms: conditions — Diabesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabesity: People with diabetes and obesity
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — It is an registry so no intervention will be used.

SUMMARY:
All participants of the Diabesity Register will receive structured assessment by nurses guided by the JADE portal at baseline including eye, feet, blood and urine examination with evaluation of BMI, blood pressure, HbA1c, lipid profile, renal and liver function tests, urine for albumin-creatinine ratio. All patients will return at 3-year for a repeat assessment of physical and psychological health, as well as changes over time.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes;
2. Obesity reaching action level as defined as body mass index (BMI) 27.5 kg/m2 and/or waist circumference (WC) 80cm in women and 90cm in men;
3. Age between 18 and 50 years;
4. Able to conversate with smartphone technology and web-based program.
5. Able to read Chinese and communicate using Chinese.

Exclusion Criteria:

1. Type 1 diabetes;
2. Active malignant disease including those with history of malignant disease less than 5 years of disease-free duration;
3. Life expectancy less than 12 months;
4. Any medical illness or condition as judged by the investigators as ineligible to participate the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All study subjects will be recruited from the Diabetes Mellitus and Endocrine Centre (DMEC) at PWH. Since 1995, the PWH runs a comprehensive complication screening program as part of a quality improvement program in the DMEC. On a weekly basis, patients with diabetes mellitus undergo comprehensive assessments for risk factors and complications by nurses and health care assistants using standard protocols.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
A composite of incidence | 3 years
  Incidence of diabetes-related complications

SECONDARY OUTCOMES:
Incidence of diabetic mellitus retinopathy | 3 years
Incidence of diabetic mellitus nephropathy | 3 years
Incidence of diabetic mellitus neuropathy | 3 years
Incidence of myocardial infarction | 3 years
Incidence of stroke | 3 years
Incidence of peripheral artery disease | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine and Therapeutics, The Chinese University of Hong Kong (CUHK), Ward 3M, Diabetes and Endocrine Research Centre, 3/F Day Treatment Block and Children Wards (Old Block), Prince of Wales Hospital, Hong Kong, Hong Kong